CLINICAL TRIAL: NCT01230658
Title: Prophylactic Enoxaparin Dosing in Roux-en-Y Gastric Bypass Surgery Patients at the St. Vincent Carmel Bariatric Center of Excellence
Brief Title: Prophylactic Enoxaparin Dosing in Roux-en-Y Gastric Bypass Surgery Patients at St. Vincent Carmel
Status: Completed | Type: Observational
Sponsor: Ascension St. Vincent Carmel Hospital (Other)
Responsible Party: Principal Investigator, Karen Wall, Pharmacist, Ascension St. Vincent Carmel Hospital
Other Study IDs: STV IRB R2009-111
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2012-11

CONDITIONS: Obesity
Keywords: prophylactic enoxaparin; Roux en Y gastric bypass surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess anti-factor Xa concentrations in patients given prophylactic enoxaparin after bariatric surgery.

DETAILED DESCRIPTION:
FDA-approved enoxaparin dosing for venous thromboembolism (VTE) prophylaxis is a fixed-dose regimen irrespective of body mass index (BMI) or actual body weight (ABW). Clinical trials suggest that dosing may be inadequate for obese patients. We plan to assess anti-factor-Xa concentrations in patients who received prophylactic enoxaparin after bariatric surgery.

This prospective study will examine 150 anti-factor Xa concentrations from patients 18 years or older undergoing primary Roux-en-Y gastric bypass surgery at St. Vincent Carmel Bariatric Center of Excellence. Patients receive varying prophylactic enoxaparin regimens at the surgeon's discretion. Anti-factor-Xa concentrations are obtained at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older undergoing primary roux-en-Y gastric bypass surgery at St. Vincent Carmel Bariatric Center of Excellence

Exclusion Criteria:

* Receiving anticoagulation therapy prior to surgery (i.e. warfarin)
* Did not receive enoxaparin after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older undergoing primary roux-en-Y gastric bypass surgery at St. Vincent Carmel Bariatric Center of Excellence.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Anti-factor Xa concentrations from patients 18 years or older undergoing primary Roux-en-Y gastric bypass surgery at St. Vincent Carmel Bariatric Center of Excellence | Anti-factor Xa concentrations obtained at steady state (3-5 hours after third enoxaparin dose)

SECONDARY OUTCOMES:
Thrombotic events - DVT confirmed by doppler guided ultrasound or PE confirmed by CT scan | within 30 days of surgery
Hemorrhagic events - defined as a change in hemoglobin greater than 3 G/dL, transfusion of packed red blood cells, endoscopic procedure indicating GI bleeding, or other major bleeding event documented by physician. | within 30 days of surgery
Re-admissions to a hospital within 30 days of surgery due to thrombotic or hemorrhagic event | within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Wall, PharmD, Principal Investigator — Ascension St. Vincent Carmel Hospital
Locations (1):
- St. Vincent Carmel Bariatric Center of Excellence, Carmel, Indiana, United States